CLINICAL TRIAL: NCT06617884
Title: Comparison of Two Home-based Gait and Balance Trainings With Different Training Frequencies in Patients With Parkinson's Disease and Ataxia
Brief Title: Home-based Gait and Balance Training in Patients With Movement Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Forschungszentrum Juelich (Other)
Collaborators: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Martina Minnerop, MD, Principal Investigator, Forschungszentrum Juelich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-1994
Record Dates: First submitted 2024-09-20; First posted 2024-10-01 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Ataxia; Parkinson Disease
Keywords: Training; home-based; video-based; motion capturing; movement disorders; Ataxia; PD; Parkinsons Disease
MeSH Terms: conditions — Ataxia; Parkinson Disease; Movement Disorders | interventions — Gait

STUDY DESIGN:
Intervention Model Description: All patients initially take part in a one-week familiarization phase without training and are then randomly assigned to one of the two training protocols or to the control group without additional training. The two different training protocols are: 20 minutes of training per day, four days per week; or 40 minutes of training per day, only two days per week. The patients who were assigned to the control group without additional training can also complete the training after the end of the study.
Who Masked: Investigator
Masking Description: The investigator who carries out the neurological examination after the training phase is blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 4 x 20 minutes training per week (Experimental): During the three-week training phase, the video-based training should be carried out at home four times a week for 20 minutes each time. The access to the training videos is provided via links.
  Interventions: Other: Gait and balance training
- 2 x 40 minutes training per week (Experimental): During the three-week training phase, the video-based training should be carried out at home two times a week for 40 minutes each time. The access to the training videos is provided via links.
  Interventions: Other: Gait and balance training
- control group (No Intervention): During the three weeks between study visit two and study visit three, no additional training is conducted. Patients who were assigned to the group without training are given access to the training material after the end of the study and can carry it out afterwards.

INTERVENTIONS:
Other: Gait and balance training — The training includes individually adapted, targeted, video-based coordination and balance training, which should lead to an improvement in gait and balance. It includes strength, coordination and flexibility exercises.
  Arms: 2 x 40 minutes training per week; 4 x 20 minutes training per week

SUMMARY:
The research project is an experimental study with three study visits at the study site at the University Hospital Düsseldorf (UKD) / Heinrich Heine University Düsseldorf (HHU) and a three-week training phase in a parallel design. Patients with movement disorders (ataxia or Parkinson's disease) can take part. The training phase includes individually adapted, targeted, video-based coordination and balance training, which should lead to an improvement in gait and balance. Two different training protocols are carried out in parallel for three weeks each: One with 20 minutes of training per day, four days per week; and one with a training duration of 40 minutes per day, only two days per week. All patients initially take part in a one-week familiarization phase without training and are then randomly assigned to one of the two training protocols or the control group without additional training. In both training phases, the total amount of weekly training time is the same, but the frequency and duration of training sessions per week differs. The patients who were assigned to the control group without additional training can complete the training after their third study visit.

DETAILED DESCRIPTION:
It will be investigated separately for the two patient groups (ataxia, Parkinsons disease), whether the video-based training can lead to an improvement in gait and balance and whether the training protocols differ with regard to the desired improvement. The gait and balance variables recorded using the two standard methods (force plate, motion capturing system) will serve as the basis for assessing the training effect. Furthermore, the investigators want to analyze how the individual variables differ between the healthy subjects (from our previous study) and patients with movement disorders.

Patients can also voluntarily record movement data using their own smartphone. This has the advantage that data can also be collected at home, which is more likely to reflect the everyday life of the participants. In particular, the aim is to check whether the data collected with the smartphone can also be read and analyzed in patients, despite the increased movement variability, and whether typical movement patterns and training-related changes can be recorded.

Only adults will take part in the study. The aim is to assess 21 patients with cerebellar ataxia or idiopathic Parkinsons disease per group. This number is based on a power calculation with the software G*Power 3.1.9.7 (Test family t tests, Means: Difference between two independent means (two groups)), with one-sided significance with α = 0.05, 1-β = 0.8 and a calculated effect size of 0.8. Participants in the study will be fully informed in advance about the study procedure. Participation in the study is voluntary. Participants can withdraw from the study at any time without giving reasons and without any disadvantages. A clinical diagnosis of cerebellar ataxia or idiopathic Parkinsons disease is a prerequisite for participation in the study. Participants must also be able to walk independently for 2 minutes. Exclusion criteria are other diseases with an impact on motor skills or serious primary psychiatric illnesses, current drug or alcohol dependency, consumptive illnesses or a poor general condition. There must be no increased risk of falling. Parkinsons patients should carry out the measurements on site and at home during the on-phase of the medication, approx. 2 hours after taking the medication. Patients are recruited via the special outpatient clinic for movement disorders at the Institute for Movement Disorders and Neuromodulation at the UKD / HHU Düsseldorf.

The study is discontinued for the individual study participant if an increased risk of falls becomes apparent. The study as a whole will be discontinued if it becomes apparent that the risks of the study outweigh the benefits or if unforeseen complications arise during the training phase.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of cerebellar ataxia or idiopathic Parkinson's syndrome
* opportunity to walk a distance of four meters unhindered at home

Exclusion Criteria:

* other diseases with an impact on motor skills
* severe primary psychiatric illnesses
* current drug or alcohol addiction
* consumptive diseases
* poor general condition
* increased risk of falling (anamnestic fall frequency of ≥ 1x per week or as assessed by the attending physician)
* incapacitated patients in official or court custody or patients unable to give consent
* for PD patients taking medication: not being able to carry out the measurement in the on-phase of the medication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-01-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
gait velocity | From enrollment to the end of intervention at 4 weeks (training groups) / at 7 weeks (control groups)
  measured in m/s, measured by a force plate (zebris), a motion capturing system (Xsens) and individual smartphones of the participants at week 0, at baseline (week 1), after training or no training (week 4) and after training for the control group (week 7).

SECONDARY OUTCOMES:
stride time | From enrollment to the end of intervention at 4 weeks (training groups) / at 7 weeks (control groups)
  time needed for one stride (two steps) measured in s, measured by a force plate (zebris), a motion capturing system (Xsens) and individual smartphones of the participants at week 0, at baseline (week 1), after training or no training (week 4) and after training for the control group (week 7).
step width | From enrollment to the end of intervention at 4 weeks (training groups) / at 7 weeks (control groups)
  measured in cm, measured by a force plate (zebris), a motion capturing system (Xsens) and individual smartphones of the participants at week 0, at baseline (week 1), after training or no training (week 4) and after training for the control group (week 7).
cadence | From enrollment to the end of intervention at 4 weeks (training groups) / at 7 weeks (control groups)
  number of steps per second, measured in s^-1, measured by a force plate (zebris), a motion capturing system (Xsens) and individual smartphones of the participants at week 0, at baseline (week 1), after training or no training (week 4) and after training for the control group (week 7).
Lat Step Dev | From enrollment to the end of intervention at 4 weeks (training groups) / at 7 weeks (control groups)
  Lateral Step Deviation / step width variability (SD / CV), measured in cm, measured by a force plate (zebris), a motion capturing system (Xsens) and individual smartphones of the participants at week 0, at baseline (week 1), after training or no training (week 4) and after training for the control group (week 7).
Toe Out Angle | From enrollment to the end of intervention at 4 weeks (training groups) / at 7 weeks (control groups)
  Foot rotation, measured in degrees, measured by a force plate (zebris) and a motion capturing system (Xsens) at week 0, at baseline (week 1), after training or no training (week 4) and after training for the control group (week 7).
Double Support Time | From enrollment to the end of intervention at 4 weeks (training groups) / at 7 weeks (control groups)
  Double Support Time, measured percentage of whole gait cycle, measured by a force plate (zebris) and a motion capturing system (Xsens) at week 0, at baseline (week 1), after training or no training (week 4) and after training for the control group (week 7).
Toe Off Angle | From enrollment to the end of intervention at 4 weeks (training groups) / at 7 weeks (control groups)
  Take off angle of foot at "toe off" position, measured in degrees, measured by a motion capturing system (Xsens) at week 0, at baseline (week 1), after training or no training (week 4) and after training for the control group (week 7).
sway area | rom enrollment to the end of intervention at 4 weeks (training groups) / at 7 weeks (control groups)
  Center of mass / center of pressure 95% ellipse area, measured in mm2, measured in all stance tasks by a force plate (zebris), a motion capturing system (Xsens) and individual smartphones of the participants at week 0, at baseline (week 1), after training or no training (week 4) and after training for the control group (week 7).
sway velocity | From enrollment to the end of intervention at 4 weeks (training groups) / at 7 weeks (control groups)
  Center of mass / center of pressure path length per time, measured in mm/s, measured in all stance tasks by a force plate (zebris), a motion capturing system (Xsens) and individual smartphones of the participants at week 0, at baseline (week 1), after training or no training (week 4) and after training for the control group (week 7).
sway path | From enrollment to the end of intervention at 4 weeks (training groups) / at 7 weeks (control groups)
  Center of mass / center of pressure path in xy-plane, measured in mm, measured in all stance tasks by a force plate (zebris), a motion capturing system (Xsens) and individual smartphones of the participants at week 0, at baseline (week 1), after training or no training (week 4) and after training for the control group (week 7).
arm-pelvis distance | From enrollment to the end of intervention at 4 weeks (training groups) / at 7 weeks (control groups)
  Distance from the arms to the pelvis, measured in mm, measured in all stance tasks by a motion capturing system (Xsens) at week 0, at baseline (week 1), after training or no training (week 4) and after training for the control group (week 7).
foot elevation | From enrollment to the end of intervention at 4 weeks (training groups) / at 7 weeks (control groups)
  maximum foot elevation during gait, measured in cm, measured in all gait tasks by a motion capturing system (Xsens) at week 0, at baseline (week 1), after training or no training (week 4) and after training for the control group (week 7).
trunk ROM | From enrollment to the end of intervention at 4 weeks (training groups) / at 7 weeks (control groups)
  Trunk range of motion in xy-plane, measured in mm, measured by a motion capturing system (Xsens) and individual smartphones of the participants at week 0, at baseline (week 1), after training or no training (week 4) and after training for the control group (week 7).
UPDRS score | From enrollment to the end of intervention at 4 weeks (training groups) / at 7 weeks (control groups)
  Unified Parkinson Disease Rating Scale, assessed via neurological examination at week 0, after training or no training (week 4) and after training for the control group (week 7), only for the patient group of Parkinsons Disease.
  A higher score means a worse outcome. Range: 0-76
Hoehn and Yahr score | From enrollment to the end of intervention at 4 weeks (training groups) / at 7 weeks (control groups)
  Hoehn and Yahr scale, assessed via neurological examination at week 0, after training or no training (week 4) and after training for the control group (week 7), only for the patient group of Parkinsons Disease.
  A higher score means worse outcome. Range: 0-5
SCAFI score | From enrollment to the end of intervention at 4 weeks (training groups) / at 7 weeks (control groups)
  Spinocerebellar Ataxia Functional Index, assessed via neurological examination at week 0, after training or no training (week 4) and after training for the control group (week 7), only for the patient group of Ataxia.
  Separate values are reportet for the 8-meter-walk-test (8MW, in seconds, higher score means worse outcome), 9-hole pegboard test (9HPT, in seconds, higher score means worse outcome) and PATA task (PATA, number of repetitions, higher score means better outcome).
FARS-ADL score | From enrollment to the end of intervention at 4 weeks (training groups) / at 7 weeks (control groups)
  Activities of daily living, Rating Scale for Friedreichs Ataxia, assessed via neurological examination at week 0, after training or no training (week 4) and after training for the control group (week 7), only for the patient group of Ataxia.
  A higher score means worse outcome. Range: 0-36.
EQ-5D-SL score | From enrollment to the end of intervention at 4 weeks (training groups) / at 7 weeks (control groups)
  Quality of life questionnaire, assessed via questionnaire at baseline (week 1), after training or no training (week 4) and after training for the control group (week 7).
  Health status is assessed in % from 0-100, a higher score means better outcome.
TUG time | From enrollment to the end of intervention at 4 weeks (training groups) / at 7 weeks (control groups)
  time to complete Timed Up and Go test, assessed via neurological examination at week 0, after training or no training (week 4) and after training for the control group (week 7).
  Measured in seconds, a higher score means a worse outcome.
FAHW score | From enrollment to the end of intervention at 4 weeks (training groups) / at 7 weeks (control groups)
  Fragebogen zum allgemeinen habituellen Wohlbefinden (general habitual well-being questionnaire), assessed via questionnaire at baseline (week 1), after training or no training (week 4) and after training for the control group (week 7).
  A higher score means better outcome.
ABC-D score | From enrollment to the end of intervention at 4 weeks (training groups) / at 7 weeks (control groups)
  German version of the Activity-Specific Balance Confidence scale, assessed via questionnaire at baseline (week 1), after training or no training (week 4) and after training for the control group (week 7).
  Measured in mean %, a higher score means a better outcome. Range: 0-100.
MSWS-12 | From enrollment to the end of intervention at 4 weeks (training groups) / at 7 weeks (control groups)
  German Version of Multiple Sclerosis Walking Scale, assessed via questionnaire at baseline (week 1), after training or no training (week 4) and after training for the control group (week 7).
  A higher score means a worse outcome. Range: 12-60.
PDQ-39 | From enrollment to the end of intervention at 4 weeks (training groups) / at 7 weeks (control groups)
  Parkinsons Disease Questionnaire, assessed via questionnaire at baseline (week 1), after training or no training (week 4) and after training for the control group (week 7), only for the patient group of Parkinsons Disease.
  A higher score means a worse outcome. Range: 0-156.
PGIC | At the end of intervention at 4 weeks (training groups) / at 7 weeks (control groups)
  Patient global impression of change (7-point Likert scale), assessed via questionnaire, after training (week 4) or after training for the control group (week 7).
  A higher score means a better outcome. Range: -3 to 3 for each item.
SARA score | From enrollment to the end of intervention at 4 weeks (training groups) / at 7 weeks (control groups)
  Scale for the Assessment and Rating of Ataxia, assessed via neurological examination at week 0, after training or no training (week 4) and after training for the control group (week 7), only for the patient group of Ataxia.
  A higher score means a worse outcome. Range: 0-40.

CONTACTS AND LOCATIONS:
Overall Officials: Martina Minnerop, PD Dr. med., Principal Investigator — Institut für Neurowissenschaften und Medizin (INM-1), Forschungszentrum Jülich GmbH
Locations (1):
- Universitätsklinikum Düsseldorf, Institut für Klinische Neurowissenschaften und Medizinische Psychologie, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
Anonymized, aggregated data can be provided upon request.

REFERENCES:
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Miyai I, Ito M, Hattori N, Mihara M, Hatakenaka M, Yagura H, Sobue G, Nishizawa M; Cerebellar Ataxia Rehabilitation Trialists Collaboration. Cerebellar ataxia rehabilitation trial in degenerative cerebellar diseases. Neurorehabil Neural Repair. 2012 Jun;26(5):515-22. doi: 10.1177/1545968311425918. Epub 2011 Dec 2. PMID 22140200